CLINICAL TRIAL: NCT04022746
Title: Multiparametric MRI and MRE Assessment of Liver Fibrosis in Patients Treated for HCC
Brief Title: An Investigational Scan (Magnetic Resonance Elastography) in Detecting Treatment Response in Patients With Advanced Liver Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2016-1113; NCI-2019-02182 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2019-07-15; First posted 2019-07-17 (Actual); Last update posted 2025-02-19 (Actual); Status verified 2025-02

CONDITIONS: Advanced Adult Hepatocellular Carcinoma; Stage III Hepatocellular Carcinoma AJCC v8; Stage IIIA Hepatocellular Carcinoma AJCC v8; Stage IIIB Hepatocellular Carcinoma AJCC v8; Stage IV Hepatocellular Carcinoma AJCC v8; Stage IVA Hepatocellular Carcinoma AJCC v8; Stage IVB Hepatocellular Carcinoma AJCC v8
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Diagnostic (MRI/MRE) (Experimental): Patients undergo standard of care MRI and MRE over 30-90 minutes within 5 days of liver biopsy before receiving any medical treatment for HCC, at 6 weeks after medical treatment for HCC, and then every 12 weeks for up to 24 months.
  Interventions: Procedure: Magnetic Resonance Elastography; Procedure: Magnetic Resonance Imaging

INTERVENTIONS:
Procedure: Magnetic Resonance Elastography — Undergo multiparametric MRI/MRE
  Other Names: MRE
Procedure: Magnetic Resonance Imaging — Undergo multiparametric MRI/MRE
  Other Names: Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR Imaging; MRI; MRI Scan; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging

SUMMARY:
This trial studies how well an investigational scan (magnetic resonance elastography [MRE]) works with standard imaging (magnetic resonance imaging [MRI]) in detecting response to treatment in patients with liver cancer that has spread to other places in the body. Diagnostic procedures, such as MRE with MRI, may make it easier for researchers to see if the treatment for liver cancer is working.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To evaluate the ability of magnetic resonance (MR) elastography (MRE) to detect changes in hepatocellular carcinoma (HCC) between baseline and after initial 6 weeks of treatment (change in MRE liver tumor stiffness compared to percent non-viable/necrotic tumor).

SECONDARY OBJECTIVES:

I. Correlate MRE imaging measurements with patient survival (overall survival and time to tumor progression) over 18 months.

II. Correlate MRE measurements with change in tumor size and enhancement on standard of care MR imaging sequences.

OUTLINE:

Patients undergo standard of care MRI and MRE over 30-90 minutes within 5 days of liver biopsy before receiving any medical treatment for HCC, at 6 weeks after medical treatment for HCC, and then every 12 weeks for up to 24 months.

ELIGIBILITY:
Inclusion Criteria:

* Liver cancer.
* Available tumor and liver parenchyma tissue (biopsy-proven HCC).
* No contraindications to MRI (such implanted ferromagnetic or pump devices, metallic fragments in eye), as indicated on our departmental MRI screening form.
* Able to undergo informed consent.
* Not pregnant.

Exclusion Criteria:

* Contraindication to MRI (including cardiac pacemaker; ferromagnetic foreign objects in the patient; metallic eye fragments; claustrophobia).
* Inability to comply with study and/or follow-up procedures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2019-06-11 (Actual); Primary Completion 2025-02-13 (Actual); Study Completion 2025-02-13 (Actual)

PRIMARY OUTCOMES:
Change in magnetic resonance elastography (MRE) liver tumor stiffness | Baseline to 6 weeks
  Imaging measurements and percent necrosis will be summarized using mean, standard deviation (SD), and range. Pearson correlation coefficient will be estimated between imaging measurements and percent necrosis.
Change in percent non-viable/necrotic tumor | Baseline to 6 weeks
  Will be determined by pathologists using follow-up biopsy/surgery samples. Imaging measurements and percent necrosis will be summarized using mean, SD, and range. Pearson correlation coefficient will be estimated between imaging measurements and percent necrosis.

SECONDARY OUTCOMES:
Overall survival | 18 months
  Cox proportional hazard model will be used to correlate imaging measurements with survival endpoints.
Time to tumor progression | 18 months
  Logistic regression model will be used to correlate imaging measurements with response status.
Change in tumor size and enhancement | Baseline to 18 months
  Will correlate MRE measurements with change in tumor size and enhancement on standard of care MR imaging sequences. Linear mixed model will be used to correlate MRE imaging measurements with other tumor characteristics (e.g. size, etc.).

CONTACTS AND LOCATIONS:
Overall Officials: Priya Bhosale, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center — http://www.mdanderson.org

DOCUMENTS (1):
  • Informed Consent Form (2022-05-17): https://cdn.clinicaltrials.gov/large-docs/46/NCT04022746/ICF_000.pdf